CLINICAL TRIAL: NCT06840197
Title: Evaluation of Rapid Diagnostic Solutions for Emerging Infectious Diseases and CBRN Threats - Mpox Virus Clinical Study in the Democratic Republic of the Congo - DiagRaMIE-Mpox Virus-DRC
Brief Title: DiagRaMIE Mpox Virus-RDC for the Diagnostic of Monkeypox
Acronym: DiagRaMIE Mpox
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: NG Biotech (Unknown); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP 2310044
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Mpox (Monkeypox); Monkeypox Virus Infection
Keywords: Mpox; Monkeypox virus; Rapid Diagnostic Test (RDT)
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vesicle, pus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NG-TestⓇ Monkeypox virus kit — Evaluation of the performance of the rapid diagnostic test (RDT) for the detection of the Mpox virus (NG-TestⓇ Monkeypox virus kit) and comparision with PCR result (reference test)

SUMMARY:
Monkeypox, caused by a virus in the Orthopoxvirus genus, is a zoonotic disease first identified in 1970 in the Democratic Republic of Congo (DRC). This infection, primarily present in Central and West Africa, has an incubation period of 6 to 21 days and initially presents with fever, headaches, muscle pain, and swollen lymph nodes. This is followed by a skin rash that evolves over 2 to 3 weeks. Lesions can spread from the face to the hands, feet, and mucous membranes, with a centrifugal distribution pattern. Diagnosis is performed using PCR, based on samples taken from lesions or cutaneous exudates, although oropharyngeal swabs may be required if skin lesions are absent.

Since May 2022, a resurgence of cases has been observed in North America, Europe, and Africa, including the DRC. As of March 2024, 94,270 cases and 178 deaths have been reported. Although less lethal than smallpox, with a mortality rate of 1% to 10% depending on the region, monkeypox remains a health threat, especially for young children and immunocompromised individuals. In response, the Commissariat à l'Énergie Atomique (CEA) and NG Biotech have developed the NG-TestⓇ Monkeypox virus rapid diagnostic test to facilitate detection. This antigenic immunochromatographic test, based on clinical samples, offers an alternative to PCR, providing rapid results without the need for costly equipment or specialized expertise. Its validation is underway for CE marking, enabling a swift response to potential health crises.

Preclinical trials have confirmed that this test detects the Mpox virus with a detection limit of 1.10⁴ pfu/mL and shows no cross-reaction with other common organisms. This clinical performance study aims to determine the effectiveness of this device using prospectively collected clinical samples. The study seeks to validate this rapid diagnostic test (RDT) and support its CE marking. Thus, this test could serve as an alternative to conventional PCR diagnostics, which require several hours to process and necessitate costly specialized equipment and expertise.

DETAILED DESCRIPTION:
The DiagRaMIE project is designed to aid in the prevention and control of emerging or re-emerging infectious diseases and to support effective responses to potential new pandemics. Its main objective is to develop rapid diagnostic immunological tests (RDTs) for priority pathogens identified by the WHO, including the Mpox virus. Recently, monkeypox (Mpox) cases have been reported concurrently in non-endemic countries (Europe and America) and endemic regions (West and Central Africa). In response, the CEA and NG Biotech have developed an RDT to help curb potential transmission. Since its deployment, the number of cases in Europe has dropped considerably, though Mpox remains a significant health concern in Africa, especially in the Democratic Republic of Congo (DRC). This clinical performance study aims to validate a reliable diagnostic tool for both ongoing and potential future Mpox epidemics.

Objectives of the Clinical Performance Study The primary goal of this clinical performance study is to prospectively assess the effectiveness of the NG-TestⓇ Monkeypox virus kit, an RDT developed by CEA and NG Biotech, in diagnosing suspected Mpox cases. The test is based on prospective immunochromatography, with this study serving to support its CE marking.

Primary Evaluation Endpoint The primary endpoint is the participant's Mpox virus infection status, determined through PCR testing using the Xpert® Mpox kit (Cepheid), which is the reference diagnostic test (Gold Standard).

Study Design This is a prospective, multicenter study aimed at validating the diagnostic accuracy of the new RDT. Participants will include symptomatic patients suspected of Mpox infection. Each participant will undergo both the reference PCR test (Xpert® Mpox kit, Cepheid) and the newly developed RDT by CEA and NG Biotech.

Target Population Patients presenting at health facilities with signs and symptoms suggestive of Mpox will be prospectively recruited by healthcare workers. After providing information about the study and obtaining consent (from either the patient or legal guardians for minors), demographic and medical data will be collected, and two samples of vesicular exudate will be taken in addition to the routine diagnostic samples. Number of subjects declared to the insurer (having signed consent): maximum 197 patients in order to have 167 evaluable patients International Research Scope This international study will take place in the Democratic Republic of Congo, specifically in regions with high disease incidence: South Kivu, Equateur, and South Ubangi. Initially, the protocol will focus on these regions. However, if outbreaks emerge elsewhere, the study may be expanded to include additional affected areas, with participants recruited from those regions as well.

Study Duration The clinical study is planned to last for six months.

ELIGIBILITY:
Inclusion Criteria:

* Any person showing signs and symptoms, vesicles, and pustules consistent with the WHO definition of suspected Mpox cases (https://www.who.int/fr/publications-detail/WHO-MPX-Surveillance-2022.3)
* Persons aged 2 years and older:
* An adult capable of providing informed consent to participate in the study
* The legal guardian(s) capable of providing informed consent for the minor's participation in the study. For minors aged 12 to 17, their assent will also be required

Exclusion Criteria:

* Refusal to participate by the individual or their legal guardian(s)
* Person not capable of giving informed consent
* Person with symptoms that appeared more than 14 days ago
* Person presenting only with macules, papules, and crusts

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any person showing signs and symptoms, vesicles, and pustules consistent with the WHO definition of suspected Mpox cases
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
To prospectively evaluate the performance of the rapid diagnostic test (RDT) for the detection of the Mpox virus (NG-TestⓇ Monkeypox virus kit), developed by the CEA and NG Biotech, based on the immunochromatography method in a prospective manner | 48 hours
  The results of the NG-TestⓇ Monkeypox virus kit will be obtained within 20 minutes (5 minutes for sampling + 15 minutes for the test) after the patient is included in the study, and these results will be compared to the PCR result, which usually requires 48 hours

CONTACTS AND LOCATIONS:
Locations (3):
- Republic of the Congo (3):
  - INRB, Mbandaka, Equateur
  - INRB, Gemena, Sud Ubangi
  - INRB, Bukavu, Sud-Kivu

IPD SHARING:
Plan to Share IPD: No